CLINICAL TRIAL: NCT06802302
Title: Effectiveness of a School-based Obesity Prevention Program on Body Fat At 6 Months of Mexican Children: a Cluster Randomized Controlled Trial
Brief Title: Effectiveness of a School-based Obesity Prevention Program on Body Fat At 6 Months of Mexican Children
Acronym: PPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Collaborators: Centro de Investigación en Alimentación y Desarrollo A.C. (Other); Instituto Nacional de Geriatria, Mexico (Other Government)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Full-time professor, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PPN2025
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Childhood Obesity Pevention
Keywords: Intervention; Nutrition; Physical activity; Randomized controlled trial; Body fat; School
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Schools that meet the inclusion/exclusion criteria will be randomly assigned to one of three groups: 1) a program implemented by nutrition and physical activity students (NUT-PA group), 2) a program delivered by physical education teachers and physical activity students (PEST-PA group), or 3) a control group.
Who Masked: Outcomes Assessor
Masking Description: A nutrition team independent of the recruitment and blinding to the study groups will carry out the measurements. The person that will do the randomly allocation of the schools will be independentof the recruitment and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NUT-PA group: intervention delivered by advanced nutrition and physical activity students. (Experimental): This group will implement the Planet Nutrition program. Advanced nutrition students will deliver one 1-hour nutrition lesson per week during school hours and will also provide nutrition and health information to parents. Additionally, advanced physical activity students will lead two 1-hour exercise sessions per week at school.
  Interventions: Behavioral: Planet Nutrition Program
- PEST-PA group: physical education schoolteachers and physical activity students. (Experimental): This group will implement the Planet Nutrition program. Advanced nutrition students will deliver one 1-hour nutrition lesson per week during school hours and will also provide nutrition and health information to parents. Additionally, advanced physical activity students will lead two 1-hour exercise sessions per week at school.
  Interventions: Behavioral: Planet Nutrition Program
- Control group (No Intervention): The schoolchildren in this group will continue with their regular nutrition and physical activity classes. At the end of the study, they will receive a printed handbook with nutrition recommendations and gain access to the materials from the Planet Nutrition program via a website.

INTERVENTIONS:
Behavioral: Planet Nutrition Program — The intervention in this study will be the same for both intervention groups, both based on the previously designed and tested "Planet Nutrition" Program (PNP). The program components include: nutrition education lessons (one 1-hour session per week), physical activity classes (two 1-hour sessions per week), and nutrition information for parents. The intervention will be implemented from February to June 2025.
  Arms: NUT-PA group: intervention delivered by advanced nutrition and physical activity students.; PEST-PA group: physical education schoolteachers and physical activity students.

SUMMARY:
School-based programs are an essential strategy for preventing obesity, yet the most effective way to implement them remains unclear. This study aims to evaluate the effectiveness of a school-based obesity prevention program, delivered by different implementers, in comparison to a control group, focusing on body fat reduction in Mexican children. This is a cluster randomized controlled trial. Approximately six public elementary schools (240 children) in Hermosillo, Mexico, will be invited to participate. Schools will be randomly assigned to one of three groups: a program implemented by advanced undergraduate students in Nutrition and Physical Activity (NUT-PA), a program implemented by Physical Education teachers and Physical Activity students (PEST-PA), or a control group. The intervention will consist of a 6-month obesity prevention program that includes nutrition education, physical activity sessions, and parent participation. The control group will continue with their regular school activities. The primary outcome will be the difference in body fat percentage at 6 months between the NUT-PA group and the control group, as well as between the PEST-PA group and the control group. Secondary outcomes will include BMI Z-score, waist circumference, and various lifestyle parameters. A mixed-effects linear analysis will be conducted using an intention-to-treat approach.

DETAILED DESCRIPTION:
This is a cluster randomized controlled trial with three parallel groups and a 1:1:1 allocation ratio. The current protocol represents the definitive phase of the study, which was previously registered and approved in clinical trials (NCT05461703). The project has been approved by the Research Ethics Committee of the Nursing Department at the Universidad de Sonora (EPD-007-2022).

ELIGIBILITY:
Schools

Inclusion Criteria:

* School principals, 4th- and 5th- grade teachers willing to participate, availability of space for physical activity classes, and groups with a minimum of 20 students.

Exclusion Criteria:

* Participating in a similar study.

Children

Inclusion Criteria:

* To be a 4th or 5th grade student (9 to 12 years) in one of the participating schools. To be eligible for this study, parents and children will be required to sign an informed consent and assent form, respectively, and had to complete anthropometric measurements (children) and lifestyle questionnaires (parents).

Exclusion Criteria:

* A personal condition that prevents conducting physical activity or a condition that parents consider should exclude their child from participating.

Implementers

Inclusion Criteria:

-Received 80% of the program training. Satisfactory response to a questionnaire that assessed their knowledge of the program following the training.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
Mean difference in body Fat (%) | At 6 months ( from baseline to the end of the study).
  Body composition will be obtained using electrical bioimpedance RJL Quantum II (Clinton Township, Michigan) following the methodology recommended by the manufacturer. With obtained data (resistance and reactance values in ohms), an equation previously designed to estimate fat-free mass in Mexican children will be used. Fat mass will be obtained by subtracting the kilograms of fat-free mass from the total kilograms of the subject and its percentage with respect to total body weight will be also calculated.

SECONDARY OUTCOMES:
Mean difference in BMI Z-score | At 6 months ( from baseline to the end of the study).
  Will be calculated using the weight, height, sex, and date of birth of the children, using the "Anthro Plus" v.1.0.4 software, which uses the WHO reference tables.
Mean difference in waist circumference | At 6 months ( from baseline to the end of the study).
  The measurement will be taken at the umbilical scar level (under the skin), with the participant standing, using a metallic anthropometric tape (Lufkin Executive Thineline W606PMM). Participants will be asked to indicate their umbilical scar location and to inhale and exhale prior to the measurement.
Difference in food consumption | At 6 months ( from baseline to the end of the study).
  Some questions from the semi-quantitative food frequency questionnaire (FFQ) from the National Health and Nutrition Survey (ENSANUT) will be used. Participants will be asked about the frequency of consumption of ultra-processed foods (sweet beverages, fried foods, cakes, and cookies) and healthy foods (fruits, vegetables, and water) in the previous 7 days. For each food, the size of the portion consumed was asked, considering an average portion established in the FFQ. Parents will answer the children's questionnaires.
Mean difference in physical activity and sedentary behavior | At 6 months ( from baseline to the end of the study).
  The questions on physical activity and sedentary lifestyle will be used from "The Health Behavior in School-Age Children" (HBSC) questionnaire. The questionnaire includes questions about the days and time (intensity, duration, and frequency) dedicated to physical activity in the last 7 days. In addition, the questionnaire includes a section on time dedicated to sedentary activities during the week and on the weekend.
Mean difference in quality of Life scores | At 6 months ( from baseline to the end of the study).
  The PedsQL™ questionnaire (Pediatric Quality of Life Inventory) will used to evaluate aspects of quality of life. This generic health status instrument assesses the frequency of problems experienced in the past month in the following aspects: physical, emotional, social, and school functioning. Responses are on a 5-point Likert scale (never = 0 to always = 4). The score for each item was inverted and converted to a linear scale from 0 to 100, with a higher score indicating a better quality of life.
Mean difference in nutrition knowledge | At 6 months ( from baseline to the end of the study).
  A questionnaire designed by the study team will be used to assess knowledge on nutrition issues. It consists of 19 questions about nutrition and health. Knowledge was evaluated on a scale from 0 to 10, with the more correct answers, the higher the score.
Feasibility of the intervention | At 6 months ( from baseline to the end of the study).
  The feasibility of the implementation of the program will be evaluated with retention, acceptability, adherence and fidelity.
  Retention: number of schools and participants that completed the final measurements.
  Acceptability: A questionnaire will be applied to children, parents, and implementers to evaluate the acceptability of the program and materials on a scale from 0 to 10.
  Adherence: number of nutrition and phisical activity classes attended by children.
  Fidelity: number of classes delivered by implementers.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Díaz Zavala, Principal Investigator — Universidad de Sonora

IPD SHARING:
Plan to Share IPD: No
Participant data (without sensitive information) may only be shared at the discretion of the principal investigator and for research purposes.

REFERENCES:
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Currie C, Inchley J, Molcho M, Lenzi M, Veselska Z, Wild F. Health Behaviour in School-Aged Children (HBSC) Study Protocol: Background , Methodology and Mandatory Items for the 2013/14 Survey.; 2014. http://www.hbsc.org
- [Background] Shamah-Levy T, Vielma-Orozco E, Heredia-Hernández O, Romero-Martínez M, Mojica-Cuevas J CNL, Santaella-Castell JA RDJ. Encuesta Nacional de Salud y Nutrición 2018-19: Resultados Nacionales.; 2020. Accessed September 4, 2020. https://ensanut.insp.mx/encuestas/ensanut2018/informes.php
- [Background] Marfell-Jones M, Olds T, Stewart A, Carter L. International Standards for Anthropometric Assessment. First edit. (ISAK, ed.).; 2006.
- [Background] Ramirez E, Valencia ME, Bourges H, Espinosa T, Moya-Camarena SY, Salazar G, Aleman-Mateo H. Body composition prediction equations based on deuterium oxide dilution method in Mexican children: a national study. Eur J Clin Nutr. 2012 Oct;66(10):1099-103. doi: 10.1038/ejcn.2012.89. Epub 2012 Jul 18. PMID 22805494
- [Background] WHO. Growth Reference 5-19 years. BMI-for-age (5-19 years). 2007. https://www.who.int/growthref/en/
- [Background] Ramírez Rivera DL, Martínez Contreras T, Villegas Valle RC, et al. Effectiveness of a school-based obesity prevention program on the BMI Z-score and body fat at 6 months in Mexican children: study protocol of a cluster randomized controlled trial. Biotecnia. 2023;25(3):71-78. doi:10.18633/biotecnia.v25i3.2074
- [Background] Ramírez-Rivera DL, Martínez-Contreras Teresita, Henry-Mejia Gricelda, et al. Efecto de una intervención en línea de cambio en el estilo de vida sobre el puntaje zIMC de escolares mexicanos: protocolo de ensayo controlado aleatorizado piloto cegado a evaluadores
- [Background] Ramirez-Rivera DL, Martinez-Contreras T, Villegas-Valle RC, Henry-Mejia G, Quizan-Plata T, Haby MM, Diaz-Zavala RG. Preliminary Results of the Planet Nutrition Program on Obesity Parameters in Mexican Schoolchildren: Pilot Single-School Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jan 18;18(2):790. doi: 10.3390/ijerph18020790. PMID 33477722
- [Background] Spiga F, Davies AL, Tomlinson E, Moore TH, Dawson S, Breheny K, Savovic J, Gao Y, Phillips SM, Hillier-Brown F, Hodder RK, Wolfenden L, Higgins JP, Summerbell CD. Interventions to prevent obesity in children aged 5 to 11 years old. Cochrane Database Syst Rev. 2024 May 20;5(5):CD015328. doi: 10.1002/14651858.CD015328.pub2. PMID 38763517
- [Background] Shamah-Levy T, Gaona-Pineda EB, Cuevas-Nasu L, et al. Prevalence of overweight and obesity in Mexican school-aged children and adolescents. Ensanut 2020-2022. Salud Publica Mex. 2023;65. doi:10.21149/14762
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in underweight and obesity from 1990 to 2022: a pooled analysis of 3663 population-representative studies with 222 million children, adolescents, and adults. Lancet. 2024 Mar 16;403(10431):1027-1050. doi: 10.1016/S0140-6736(23)02750-2. Epub 2024 Feb 29. PMID 38432237